CLINICAL TRIAL: NCT02615522
Title: Prospektive, Klinische Verlaufsuntersuchung (Post Market Follow-Up) Der primären Knieendoprothese BPK-S Integration
Brief Title: Prospective Post Market Clinical Follow-Up of the Primary Knee Endoprosthesis BPK-S Integration
Status: Terminated | Type: Observational
Sponsor: Peter Brehm GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-02-BPK-S Integration
Record Dates: First submitted 2015-11-20; First posted 2015-11-26 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee; Joint Instability
Keywords: primary TKR
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Instability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BPK-S Integration

SUMMARY:
Prospective, monocenter post market clinical follow-up of a primary knee replacement bearing the CE-mark.

200 subjects will be recruited and followed up for up to ten years or until revision of the primary knee endoprosthesis, whichever occurs first. Documentation of clinical and radiological parameters within the clinical routine pre-operative and post-operative at 3 and 12 months and 2, 5 and 10 years to evaluate time to revision, pain situation, knee functionality, mobility and stability.

ELIGIBILITY:
Inclusion Criteria:

* Congenital or acquired knee joint defects/deformation or
* Defects or malfunction of the knee joint or
* Arthrosis (degenerative, rheumatic) or
* Post-traumatic arthritis or
* Symptomatic knee instability or
* Reconstruction of flexibility or
* Patients with metal hypersensitivity (ceramic tibia/femur)

Exclusion Criteria:

* Illnesses which can be treated without using a knee joint implant.
* Acute or chronic infections near the implantation
* Systemic diseases and metabolic disorders
* Serious osteoporosis
* Serious damage to the bone structures that impedes stable implantation of the implant components
* Diseases that impair bone growth, e.g. cancer, renal dialysis, osteopenia, etc.
* Bone tumors in the area of the implant anchoring
* Obesity or overweight of the patient
* Overload of the knee implant to be expected
* Abuse of medication, drug abuse, alcoholism or mental disease
* Lack of patient cooperation
* Sensitivity to foreign matter in the implant materials
* Patients under the age of 18
* Patients participating in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary total knee endoprosthesis with BPK-S Integration of age 18 and older
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Time until revision | 10 years

SECONDARY OUTCOMES:
Improvement of clinical situation based on Knee Society Score | 3 and 12 months, 2, 5, 10 years
Documentation of incidents | Up to 10 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Landesklinikum Amstetten, Amstetten, Lower Austria, Austria